CLINICAL TRIAL: NCT06463327
Title: An Open-label, Multicenter, Phase 1 Study to Evaluate Safety and Preliminary Efficacy of Intravenous TCB008 in Patients With Relapse or Refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)/AML
Brief Title: ACHIEVE2 - Safety and Preliminary Efficacy of Intravenous TCB008 in Patients With Relapse or Refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)/AML
Acronym: ACHIEVE2
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TC Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCB008-003
Record Dates: First submitted 2024-05-08; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Receptors, Antigen, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Drug product: TCB008 Administration route: Intravenous infusion
  Proposed Dose Limits (DL) for dose escalation:
  * Cohort 1: 1.5 mL IV TCB008 (3.6×107 to 6.9×107 cells)
  * Cohort 2: up to 5 mL IV TCB008 (12.0×107 to 23.0×107 cells)
  * Cohort 3: up to 18 mL IV TCB008 (43.2×107 to 82.8×107 cells)
  The DL for the dose expansion will be based on the recommended dose for expansion determined in the dose escalation part of the study
  Dosing is intended to be fixed (i.e., not weight-based or body surface area-based).
  In both the dose escalation and dose expansion parts of the study, participants may be reinfused with TCB008 up to 3 times following initial infusion, if deemed appropriate by the investigator (or designee) based on review of available safety data and confirmation of disease status.
  In the case that TCB008 is reinfused each dose will be administered 29 days apart.
  Interventions: Drug: TCB008

INTERVENTIONS:
Drug: TCB008 — TCB008 is derived from the peripheral blood mononuclear cells (PBMCs) of unrelated, healthy donors and consists of expanded cluster designation (CD)3+ T cells expressing the γ chain variable region 9 δ-chain variable region 2 (Vγ9Vδ2) T cell receptor (TCR); it is infused into patients to boost their immune system. It is currently developed for treatment of cancers and infectious diseases.
  Other Names: CD3+ T cells expressing the γ-chain variable region 9 δ-chain variable region 2 (Vγ9Vδ2) T cell receptor (TCR)

SUMMARY:
TCB008-003 (ACHIEVE2) is an open-label, multi-center study conducted in 2 parts (dose escalation followed by dose expansion) to evaluate safety, persistence/expansion, and preliminary efficacy of single and multiple intravenous doses of TCB008 in patients with Relapse or Refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)/AML, who have failed or are intolerant to the current standard of care. The dose escalation will follow a 3+3 design with 3 cohorts planned. Once the recommended dose for further investigation has been confirmed, based on dose-limiting toxicities (DLTs), overall safety data, and preliminary efficacy data, up to 20 patients will be enrolled to into one of each of the three dose expansion cohorts.

DETAILED DESCRIPTION:
TCB008-003 (ACHIEVE2) is an open-label, multi center study conducted in 2 parts (dose escalation followed by dose expansion). The purpose of this study is to evaluate Safety and Preliminary Efficacy of Intravenous TCB008 in Patients with Relapse or Refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)/AML.

TCB008 is derived from the peripheral blood mononuclear cells (PBMCs) of unrelated, healthy donors and consists of expanded cluster designation (CD)3+ T cells expressing the γ-chain variable region 9 δ-chain variable region 2 (Vγ9Vδ2) T cell receptor (TCR); it is infused into patients to boost their immune system. It is currently developed for treatment of cancers and infectious diseases.

Approximately 69 people will take part in this study at several different locations throughout the United States of America.

In both parts of the study, potential patients will be screened to assess their eligibility to enter the study within 35 days prior to the first dose of the investigational medicinal product (IMP). Once enrolled in the study patients will undergo lymphodepletion chemotherapy prior to administration of the IMP using the following regimen: fludarabine (30 mg/m2/day) will be administered from Days -6 to -3 (total 120 mg/m2), cyclophosphamide (0.5 g/m2/day) from Days -5 to -3 (total 1.5 g/m2), followed by 2 days of rest (Days -2 and -1).

The dose escalation part will use a 3+3 design.

The dose escalation part will comprise 3 cohorts of 3 to 6 patients where patients in each cohort will receive up to 4 doses of TCB008 in accordance to the cohort to which they are assigned (initial infusion plus 3 potential reinfusions) with the following dose-level (DL) escalating for each cohort:

Cohort 1: 1.5 mL IV TCB008 (3.6×107 to 6.9×107 cells) Cohort 2: up to 5 mL IV TCB008 (12.0×107 to 23.0×107 cells) Cohort 3: up to 18 mL IV TCB008 (43.2×107to 82.8×107 cells)

Decisions to escalate the dose will be made on any observed DLTs as well as additional supportive data such as overall safety profile from the 28-day DLT evaluation period following the first infusion with TCB008 for all patients of a cohort. The Safety Review Committee (SRC; with agreement from the sponsor [or designee]) may elect to pursue intermediate, lower, or higher DLs based on overall review of safety data. Alternative dosing schedules may also be considered based on the emerging safety data.

The dose expansion part will start once dose escalation has been completed. Once the recommended dose for expansion (RDE) has been confirmed, up to 20 patients will be enrolled into one of each of the following dose expansion cohorts:

Cohort 4: Patients with relapsed or refractory AML or MDS/AML Cohort 5: Patients with previously treated AML or MDS/AML who achieved in their last treatment CR with MRD Cohort 6: Patients with previously treated relapse or refractory adverse risk AML or MDS/AML per ELN guidelines 2022.

For both parts (dose escalation and dose expansion), patients may be reinfused with TCB008 up to 3 times following initial infusion (at the same dose as the initial infusion), if deemed appropriate by the investigator (or designee), based on review of available safety data and confirmation of disease status as defined below:

* CR was not achieved (AML patients) following the first dose of TCB008
* CR was achieved but MRD is present (MRD+ patients) following the first dose of TCB008
* patients' disease did not progress following administration of previous doses of TCB008.

Such reinfusions will not be preceded by lymphodepletion chemotherapy.

For both parts (dose escalation and dose expansion), the study will be conducted as follows:

* screening period: Approximately 4 weeks
* lymphodepletion chemotherapy period (right before Cycle 1): Approximately 1 week
* treatment period: Up to 16 weeks from the first dose of IMP (TCB008)
* follow-up period: Approximately 24 months from the last dose of IMP (TCB008).

Patients will be monitored for safety, tolerability, persistence/expansion, and preliminary efficacy throughout the study. Tumor response will be assessed according to ELN 2022 guidelines, 28days after the initial infusion, and second, third, and fourth reinfusions (as applicable), and starting at 6 months (±7 days), approximately every 3 months (±7 days) during the follow-up period. Optional disease assessment may be performed at the investigator (or designee)'s discretion, 14 days after the initial infusion, and second, third, and fourth reinfusions (as applicable).

Patients who discontinue treatment due to other reasons than disease progression will continue with cancer assessments as per protocol until disease progression, patient refusal, death, or starting a new anticancer treatment. The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all the following criteria at the screening visit unless otherwise stated:

1. Male or female ≥18 years of age at the time of signing the ICF
2. Body weight ≥50 kg
3. Male patients and female patients of childbearing potential will agree to abide by the contraception requirements defined in the protocol
4. Diagnosis of primary AML, AML with myelodysplasia-related changes, or MDS/AML (10% to 19% blasts in BM or peripheral blood) according to World Health Organization23 classification as determined by pathology review at the treating institution
5. Patients with AML who have relapsed or have refractory disease after at least one prior line of therapy and for whom there are no standard-of-care options, such that patients meet 1 of the following criteria (a to c) in the escalation part of the study or specified criteria for each cohort in the expansion part of the study:

   1. Refractory disease not achieving CR, CRh, or CRi after at least 2 courses of intensive induction treatment or after a defined response landmark for less intensive treatments (Cohort 4 and Cohort 6 [only patients with adverse risk per ELN guidelines 202223] for the expansion part of the study)
   2. Relapsed disease within 1 year after achieving CR, CRh, or CRi, where relapse is defined as 5% or more BM blasts that are not attributable to any other cause, reappearance of blasts in the blood in at least 2 peripheral blood samples collected at least one week apart, or development of extramedullary disease (Cohort 4 and Cohort 6 [only patients with adverse risk per ELN guidelines 202223] for the expansion part of the study)
   3. Previous treated AML or MDS/AML that achieves CR with MRD+ (Cohort 5 for the expansion part of the study)
6. Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 2
7. Adequate coagulation, defined as activated partial thromboplastin time and prothrombin time or international normalized ratio ≤1.5 × upper limit of normal (ULN)
8. Adequate hepatic function, defined as:

   1. alanine aminotransferase or aspartate aminotransferase ≤2.5 × ULN or ≤5 × ULN with documented liver involvement
   2. total bilirubin ≤1.5 × ULN or ≤3 × ULN with documented liver involvement. If total bilirubin is >1.5 × ULN then direct/indirect or conjugated/unconjugated bilirubin tests should be performed and meet the parameter specified. For patients with hemolysis and/or Gilbert's syndrome, they may be enrolled if unconjugated/indirect bilirubin is <5 × ULN.
9. Adequate renal function defined by serum creatinine up to 1.5 × ULN.
10. Cardiac left ventricular ejection fraction ≥45% and no evidence of pericardial effusion
11. Blood oxygen saturation (SaO2) >92% on room air
12. Serum albumin ≥3.0 g/dL
13. Ability to receive lymphodepletion therapy, IV infusions of IMP, comply with required assessments, including required clinic visits for the duration of study participation.
14. Adequate hematologic status within 7 days prior to the start of lymphodepletion (Day 6);

    1. platelet count ≥50×109/L, may be supported by transfusion
    2. hemoglobin ≥ 8 mg/dL, may be supported by transfusion
    3. white blood cell count ≤30×109/L, hydroxyurea may be used to achieve this level.
15. Patients must be, in the investigator (or designee)'s judgment, able and willing to comply with the study protocol.

For Patients in the Dose Escalation after the DLT Assessment:

No hematologic parameters apply but the patient must be responsive to transfusion support if given for thrombocytopenia or anemia.

Exclusion Criteria:

Patients will be excluded from the study if they satisfy any of the following criteria, as applicable, at screening unless otherwise stated:

Medical Conditions

1. Major surgery within 4 weeks prior to the planned start of lymphodepletion
2. Patients with a history of symptomatic deep vein thrombosis or pulmonary embolism requiring anticoagulation therapy within 6 months prior to enrollment
3. Hypersensitivity to iron-dextran, murine antibodies, or any of the agents used in this study
4. History of allogeneic or autologous SCT or any other organ transplant or chimeric antigen receptor-modified T cell therapy within the 60 days prior to the start of lymphodepletion (Day 6) or with any of the following:

   1. active GVHD of any grade
   2. need for anticytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity >CTCAE Grade 1 from CAR-T therapy
   3. ongoing immunosuppressive therapy.
5. Clinically active central nervous system leukemia or prior history of CTCAE Grade ≥3 drug-related central nervous system toxicity
6. Evidence of moderate to severe forms of primary immunodeficiencies. Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura) where it is required to introduce new therapy or escalate concomitant therapy within the 4 weeks prior to the start of lymphodepletion (Day 6) in order to maintain adequate blood counts
7. History of autoimmune disease resulting in significant end-organ disease or requiring systemic immunosuppression and/or systemic disease-modifying agents within the last 1 year:

   1. patients who receive a physiologic dose of steroid (prednisolone [or equivalent] 7.5mg/day or equivalent) are eligible for study participation
   2. patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for study participation
   3. patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for study participation
   4. patients with a history of immune thrombocytopenic purpura or autoimmune hemolytic anemia not requiring active treatment are be eligible.
8. Clinically significant, uncontrolled cardiac, cardiovascular disease or history of myocardial infarction, cardiac angioplasty or stenting, unstable angina, serious cardiac arrhythmia, or other clinically significant cardiac disease within 6 months prior to the first dose of IMP (TCB008), or prolongation of the QT interval corrected for heart rate (QTcF) >470 msec on all 3 consecutive electrocardiograms (ECGs) during screening

   a. correction of suspected drug-induced QTcF prolongation can be attempted at the investigator (or designee)'s discretion, only if clinically safe to do so, with either discontinuation of the offending drug or by switching to another drug not known to be associated with QTcF prolongation.
9. Significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including the below:

   1. active pulmonary disease (such as severe obstructive pulmonary disease, idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis). History of limited radiation pneumonitis is allowed.
   2. clinically significant liver disease (including cirrhosis)
   3. clinically significant neurological disease (such as cerebrovascular ischemia/hemorrhage within 6 months, dementia, seizure disorder, or cerebellar disease).
10. Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator (or designee) and the sponsor (or designee) makes it undesirable for the patient to participate in the study. Screening for chronic conditions is not required.

    a. Prophylactic antimicrobials are allowed.
11. History of infection with any of the following: HIV; hepatitis B virus (HBV), as determined by positivity for hepatitis B surface antigen or hepatitis B core antibody; or hepatitis C virus (HCV), as determined by positivity for anti-HCV antibody

    1. a history of infection with HBV or HCV may be acceptable if viral load is undetectable per qPCR and/or nucleic acid testing
    2. for patients with unknown HIV status, HIV testing will be performed at screening and the result should be negative for enrollment.
12. Previous reactions to fludarabine or cyclophosphamide or patients at risk of fludarabine related neurotoxicity
13. Acute promyelocytic leukemia
14. BCR-ABL-positive leukemia.
15. Active second malignancy unless in remission and with life expectancy >2 years, examples of allowed second malignancies include:

    1. history of malignancy that has been treated with curative intent at least 2 years prior to screening and with no evidence of relapse, if no concurrent anticancer therapy (except hormonal therapy) is being given
    2. history of malignancy with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
    3. prostate cancer with no evidence of metastatic disease and not requiring active therapy, except antiandrogen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recommended Dose of TCB008 for Dose-Expansion | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  To establish the recommended dose for further investigation in the dose-expansion part of the study, in patients with relapsed or relapsed refractory AML or MDS/AML, or MRD persistent-AML or MDS/AML (dose escalation part only).
Safety and Tolerability of TCB008 | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Incidence and severity of dose-limiting toxicities (DLTs).
  The severity grade will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. Cytokine release syndrome and neurotoxicity will be graded per American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Safety and Tolerability of TCB008 | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs). Severity of all AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Preliminary Antitumor Activity of TCB008 | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Preliminary antitumor activity of TCB008 will be determined according to European Leukemia Net 2022 Diagnosis and Management of Acute Myeloid Leukemia guidelines.

OTHER OUTCOMES:
Expansion and Persistence of γδ T cells in Peripheral Blood and/or Bone Marrow | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  This will be measured through concentrations of γδ T cells in the peripheral blood and bone marrow.
Evaluate Measurable Residual Disease (MRD) during and after therapy with TCB008 | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Characterization of the presence of AML blasts in bone marrow and/or peripheral blood, as determined by next-generation sequencing or flow cytometry methodologies.
Immunogenicity of TCB008 | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Measured through the development of anti-TCB008 antibodies.
Chimerism of allogeneic γδ T cells in peripheral blood and/or bone marrow | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Measured by Human Leukocyte Antigen (HLA) mismatch between donor and patient T cells found in blood and bone marrow samples.
Cytokine release profile of allogeneic γδ T cells in peripheral blood and/or bone marrow | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Measured by cytokine profiling in serum.
Phenotype of allogeneic γδ T cells in peripheral blood and/or bone marrow | The total duration of study participation for each patient (from screening through end of study visit) is anticipated to be approximately 29 months
  Immunophenotyping of T cells (pre- and post-infusion).

IPD SHARING:
Plan to Share IPD: Undecided